CLINICAL TRIAL: NCT04715529
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Dose-escalation and Food Effect Study to Assess the Safety, Tolerance, and Pharmacokinetics of FZJ-003 In Healthy Volunteers
Brief Title: Phase 1 Study to Evaluate Safety and Pharmacokinetics of FZJ-003 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F0025-101
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: SAD and MAD: 6 cohorts, 8 subjects take FZJ-003 and 2 subjects take placebo; Food Effect on Phamocokinetics: 14 subjects, crossover designing
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FZJ-003 (Experimental)
  Interventions: Drug: FZJ-003
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FZJ-003 — Subjects will receive FZJ-003 oral capsules in a dose escalation format.
  Arms: FZJ-003
Drug: Placebo — Subjects will receive placebo oral capsules (matching FZJ-003) in a dose escalation format .
  Arms: Placebo

SUMMARY:
A randomized, double-blinding, dose-escalated phase 1 trial to evaluate the tolerance and fasting/postprandial pharmacokinetics of FZJ-003, an oral Janus kinase1 (JAK1) inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent；
2. Communicate well with the researcher and be able to complete the research in accordance with the research regulations；
3. No plan for pregnancy in the next 6 months and voluntarily take effective contraceptive measures; No plan for sperm or egg donation；
4. Healthy male and/or female subjects between the ages of 18 and 50 years ( inclusive)；
5. Male body weight≥50.0kg or female body weight≥45.0kg; Body Mass Index (BMI) between 18 to 28 (both inclusive), calculated as weight in kg / height in m2.

Exclusion Criteria:

1. Someone smoking more than 5 pieces per day within the 3 months before the trial；
2. Suspected of being allergic to investigational drug or any ingredient in the investigational drug, or people with allergies (multi-drug or food allergies)；
3. Having a history of alcohol abuse (14 units of alcohol per week: 1 units = beer 285 mL, or 25 mL of spirits, or 100 mL of wine);
4. Blood donation or extensive blood loss ≥400 mL within 3 months before screening, or planning blood donors during the study;
5. Urine drug test positive or have a history of drug abuse or drug use in the past 5 years;
6. Subjects who were intolerant of high-fat meals (2 boiled eggs, 1 slices of buttered bacon toast, a box of fries, and a glass of whole milk) were applied only to subjects who participated in the postprandial test;
7. Taked any drug within 14 days before screening, including prescription drugs, over-the-counter drugs, Chinese herbal medicines and health products (except regular supplementary vitamins);
8. Taked any drug that changes liver drug enzyme activity within 28 days before screening, such as CYP3A4 inhibitors or inducers;
9. Major changes in diet or exercise habits within 2 weeks before screening or during the period from screening to administration;
10. Took a special diet (including dragon fruit, mango, grapefruit, etc.) or strenuous exercise, and other activities that affect drug absorption, distribution, metabolism, excretion and so on within 2 weeks before screening;
11. Received or planned to receive any vaccine within 30 days before and after the trial;
12. Participated in clinical trials within 3 months before the first administration of the study, or planned to participate in other clinical trials during the study period;
13. Having difficulty of swallowing or any history of gastrointestinal diseases that affect drug absorption;
14. With low immune function or immunodeficiency, or long-term use of immunosuppressive drugs; or used immunosuppressive drugs within 30 days before screeing;
15. Have or have had malignant tumors；
16. Active tuberculosis; or have a history of tuberculosis or latent tuberculosis infection; tuberculosis infection T cell spot test positive;
17. Any infection that has been determined to be clinically significant by the investigator within 3 months or any infection within 7 days before the study;
18. Herpes or varicella within 3 months before the trial;
19. Underwent major trauma or major surgery in 3 months before screening, or have plan for surgery in trial;
20. Have a history of diverticulitis, peptic ulcer or perforation of digestive tract；
21. Clinical laboratory tests are abnormal and have clinical significance, or other clinical findings showing clinically significant diseases (including but not limited to heart Cerebrovascular, gastrointestinal, lungs, endocrine, renal, nerves, blood, immunizations, or mental disease);
22. Active viral hepatitis (B or C) as demonstrated by positive serology at Screening；or test positive for human immunodeficiency virus (HIV) at Screening; or syphilis treponema pallidum antibody and syphilis rapid plasma reagin test are positive;
23. QTcB interval greater than (>) 470 (male) or 480 (female) milliseconds;
24. Female subjects are in lactation or serum pregnancy test are positive during screening or during the test;
25. Acute illness or combination therapy from the screening stage to administration;
26. Taking chocolate, any caffeine, or xanthine-rich food or drink at least 48 hours prior to the use of the study drug;
27. Taking any alcoholic products within 24 hours prior to the use of the study drug, or cannot limit alcohol drinks as required in trial;
28. Other circumstances that is deemed not appropriate for the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Adverse events and the number of volunteers with adverse events as a measure of safety and tolerability | up to 72 hours postdose
  Tests will be performed to assess whether the study drug has any potentially adverse effect (laboratory tests on blood and urine for functioning of organs; ECG testing). Also, participants will carefully be monitored by medical staff for vital signs, and asked to report any side effect experienced in the course of the study.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | up to 72 hours postdose
Area under the plasma concentration-time curve (AUC) | up to 72 hours postdose
Pharmacodynamics (PD) parameters of percent and actual change from baseline for a panel of JAK-dependent biomarkers | up to 24 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- the First Bethune Hospital of Jilin University, Changchun, Jilin, China